CLINICAL TRIAL: NCT00533962
Title: Anterior Juxtascleral Depot of Anecortave Acetate: Intraocular Pressure Reduction in Glaucoma Patients
Brief Title: IOP Reduction After Anecortave Acetate Injection in Glaucoma Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Collaborators: Alcon Research (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-01
Record Dates: First submitted 2007-09-20; First posted 2007-09-24 (Estimated); Last update posted 2007-09-24 (Estimated); Status verified 2007-09

CONDITIONS: Glaucoma; Intraocular Pressure
Keywords: Glaucoma; Anecortave Acetate; Intraocular pressure; Advanced glaucoma cases with uncontrolled IOP
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Anterior Juxtascleral Depot of Anecortave Acetate

SUMMARY:
Introduction: Ocular administration of glucocorticoids is a common and effective treatment for several ocular diseases. However it is often complicated with the elevation of intraocular pressure (IOP). Anecortave acetate (AA) is an analog of cortisol acetate and lacks the typical anti-inflammatory and immunosuppressive properties of glucocorticoids. The effect of its anterior juxtascleral depot (AJD) injection has been evaluated in cases of glaucoma caused by intravitreal triamcinolone acetonide, presenting impressive results. The purpose of this study is to evaluate the efficacy and safety of the AA injection as a possible antiglaucoma treatment alternative. Methods: A prospective clinical study will be carried out including 30 glaucoma patients (30 eyes). After inclusion each patient will receive a single AJD injection of 30 mg of AA in the selected eye. Main outcome measure include: intraocular pressure at 1st day, 7th day, 1st, 2nd and 3rd months.

ELIGIBILITY:
Inclusion Criteria:

* Advanced glaucoma cases with surgery or cyclophotocoagulation indication (IOP over 25 mmHg)
* Patients should be under maximum tolerated medication
* Low best corrected visual acuity (worse than 20/100)

Exclusion Criteria:

* Under 18 or over 80

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-08

PRIMARY OUTCOMES:
Intraocular pressure | Procedure

SECONDARY OUTCOMES:
Visual Acuity; side effects (biomicroscopy exam) | Post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Tiago Prata, Study Director — Federal University of São Paulo
Locations (1):
- São Paulo, São Paulo, São Paulo, Brazil